CLINICAL TRIAL: NCT02443350
Title: Multicenter and Prospective Clinical Registry Study of Anti-N-methyl-D-aspartate Receptor Encephalitis in Beijing Area
Acronym: MuPRaNE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jia Wei Wang,MD (Other)
Responsible Party: Sponsor-Investigator, Jia Wei Wang,MD, M.D.;The head of Department of Neurology and Medical Research Center, Beijing Tongren Hospital
Organization: Beijing Tongren Hospital (Other)
Other Study IDs: CH 201411101
Record Dates: First submitted 2015-05-10; First posted 2015-05-13 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Anti-N-Methyl-D-Aspartate Receptor Encephalitis
MeSH Terms: conditions — Anti-N-Methyl-D-Aspartate Receptor Encephalitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months

SUMMARY:
Anti N-methyl-D-aspartate receptor encephalitis is an autoimmune encephalitis，found in recent years，producing the specific IgG antibody induced by the NMDA receptors.It is the most common curable disease among the non infectious-autoimmune encephalitis,usually has been misdiagnosed as other causes of encephalitis.Our previous study found that there are differences between the Chinese and the foreign in anti-NMDA receptor encephalitis such as the sex ratio, the rate of combined tumor and clinical manifestations.As a new found disease,the incidence rate has been underestimated.Therefore,to establish the Registry Research Database for Chinese group of anti-NMDA receptor encephalitis is imminent.This study will combine Beijing area's hospitals and foreign experts,depending on multicenter, prospective and registry method,to understand the incidence in Beijing area,to summarize and analyze the clinical data of patients.So,there will make a solid foundation for the subsequent Beijing area detection platform and other research.

ELIGIBILITY:
Inclusion Criteria:

* Older than 6 months.
* Encephalopathy symptoms (change of mental state and consciousness level) persist for more than 24 hours;
* At least one or more clinical features of the followings: fever, epilepsy, focal neurological deficiency symptoms, changes in CSF(cerebrospinal fluid inflammatory), changes in EEG (electroencephalogram), radiographic abnormalities;
* Clinical suspected encephalitis, but conventional detected methods cannot make etiology clear

Exclusion Criteria:

* Infants less than 6 months;
* The metabolic encephalopathy;
* Infectious encephalitis with clinically clear pathogen, referring the specific pathogenic microorganisms, including: bacteria, virus, fungus, parasite, spirochete and so on;
* Non-infectious encephalitis with clinically clear diagnosis, including: multiple sclerosis, optic neuromyelitis, acute disseminated encephalomyelitis and so on.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The unexplained encephalitis patients in Beijing area
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-06; Primary Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
death | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital,Capital Medical Universiy, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Peng Y, Dai F, Liu L, Chen W, Yan H, Liu A, Zhang X, Wang X, He J, Li Y, Li C, Chen L, Zhao Y, Li L, Ma Q, Wang J. Validation of the NEOS score in Chinese patients with anti-NMDAR encephalitis. Neurol Neuroimmunol Neuroinflamm. 2020 Aug 5;7(5):e860. doi: 10.1212/NXI.0000000000000860. Print 2020 Sep. PMID 32759178